CLINICAL TRIAL: NCT06593743
Title: Proof of Concept Study in Healthy Volunteers to Investigate the Safety and Dose Response to a Single Dose (0.3%,1% or 3%) of Methoxamine (NRL001)applied to the Anus
Brief Title: The Safety and Dose Response to Single Anal Doses of NRL001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: NRL001-01/2002 (HV)
Record Dates: First submitted 2015-06-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Faecal Incontinence
MeSH Terms: conditions — Encopresis | interventions — Suppositories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (4):
- Perianal NRL001 Gel 3 strengths (Experimental): A single peri-anal application of NRL001 0.3%, 1%, 3% gel in stepwise dose ascending fashion.
  Interventions: Drug: Perianal NRL001 Gel 3 strengths
- Intraanal NRL001 Gel 2 strengths (Experimental): A single intra-anal application of 3% or 1% NRL001 gel.
  Interventions: Drug: Intraanal NRL001 Gel 2 strengths
- Intrarectal NRL001 Gel (Experimental): A single intra-rectal application of 1% NRL001 gel.
  Interventions: Drug: Intrarectal NRL001 Gel
- NRL001: 10mg suppository (Experimental): One 10mg NRL001 suppository applied to rectum.
  Interventions: Drug: NRL001: 10mg suppository

INTERVENTIONS:
Drug: Perianal NRL001 Gel 3 strengths — A single application of 0.3%, 1.0%, 3.0% NRL001 gel in stepwise dose ascending fashion.
  Other Names: methoxamine gel 0.3%, 1.0%, 3.0%
  Arms: Perianal NRL001 Gel 3 strengths
Drug: Intraanal NRL001 Gel 2 strengths — A single application of 3.0% or 1.0% Gel
  Other Names: methoxamine gel 3.0%, 1.0%
  Arms: Intraanal NRL001 Gel 2 strengths
Drug: Intrarectal NRL001 Gel — A single application of 1.0% Gel
  Other Names: methoxamine gel 1.0%
  Arms: Intrarectal NRL001 Gel
Drug: NRL001: 10mg suppository — NRL001 10mg suppository applied to rectum.
  Other Names: methoxamine suppository
  Arms: NRL001: 10mg suppository

SUMMARY:
Single centre dose-finding and proof-of-concept study in healthy volunteers to assess the effects of single doses of NRL001 on the mean anal resting pressure (MARP). In addition, the pharmacokinetics of NRL001 and subject safety are also examined.

DETAILED DESCRIPTION:
This is a single centre dose-finding and proof-of-concept study in healthy volunteers to assess the effects of single doses of NRL001 on the mean anal resting pressure (MARP). In addition, the pharmacokinetics of NRL001 and subject safety are also examined.

The study consists of four parts, which evaluate different NRL001 concentrations and sites of application. Treatments consist of a single local application of either 0.3%, 1% or 3% w/w NRL001 gel applied peri-anally, of either 1% or 3% w/w NRL001 gel applied intra-anally, or 1% w/w NRL001 administered rectally. In addition, a 10 mg NRL001-containing suppository applied to the rectum is assessed.

ELIGIBILITY:
Inclusion Criteria:

* No previous history of ano-rectal conditions/diseases.
* No history of heart disease.
* 18 to 75 years of age.
* Males and females but pre-menopausal females of child bearing potential must be using adequate contraceptive methods and have a negative pregnancy test before the start of the study.

Exclusion Criteria:

* Use of medication in the last 30 days with vasodilatory activity.
* Use of any medication in the last 30 days applied to the anus and/or via the rectum (exception: participation in Part A, Part B or Part C of NRL001-01/2002(HV)
* Regular intake of more than 21 units of alcohol per week.
* Pregnant females.
* Breast feeding mothers.
* Presence of concomitant gastrointestinal diseases or disorders, such as significant abdominal symptoms and haemorrhoids but also any significant organ (e.g. renal, hepatic or cardiac)dysfunction.
* Volunteers whom the investigator feels would not be compliant with the requirements of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-12; Primary Completion 2004-07 (Actual); Study Completion 2013-11-12 (Actual)

PRIMARY OUTCOMES:
Mean anal resting pressure | Six hours at visit 2
  Mean anal resting pressure (MARP) was recorded using anal manometric catheter

SECONDARY OUTCOMES:
Blood pressure (mmHg) | Six hours at visit 2
  Blood pressure was measured before the application of the trial medication and then every 30 minutes for the first 2 hours after application, plus 2 hourly for the remaining follow-up period.
Pulse rate (beats per minute) | Six hours at visit 2
  Pulse rate was measured before the application of the trial medication and then every 30 minutes for the first 2 hours after application, plus 2 hourly for the remaining follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine; John H Scholefield, MD, Principal Investigator — University Hospital - Queens Medical Centre
Locations (1):
- University Hospital - Queens Medical Centre, Nottingham, United Kingdom